CLINICAL TRIAL: NCT03232320
Title: A Prospective, Randomized, Multi-center, Phase III, Double-blind, Placebo-Controlled, Parallel-Group Study to Evaluate the Efficacy and Safety of MEDITOXIN in Treatment of Cervical Dystonia
Brief Title: Meditoxin® Treatment in Patients With Cervical Dystonia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Medy-Tox (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MT01-KR16CVD309
Record Dates: First submitted 2017-07-25; First posted 2017-07-27 (Actual); Last update posted 2019-03-27 (Actual); Status verified 2019-03

CONDITIONS: Dystonia; Dystonic Disorder
MeSH Terms: conditions — Dystonia; Dystonic Disorders | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MEDITOXIN (Experimental)
  Interventions: Drug: Meditoxin
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Meditoxin — Meditoxin (Botulinum toxin type A)
  Arms: MEDITOXIN
Drug: Placebo — Placebo (Normal saline)
  Arms: Placebo

SUMMARY:
To determine the efficacy and safety of Meditoxin in subjects with cervical dystonia compared with placebo (normal saline)

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 20 to less than 75 years
* Subjects requiring treatment for a clinical diagnosis of cervical dystonia with Toronto Western Spasmodic Torticollis Rating Scale(TWSTRS)-Total Score >=20 and TWSTRS-Severity score >=10

Exclusion Criteria:

* Subjects with pure anterocollis
* Subjects with neuromuscular junctional disorders (e.g., myasthenia gravis, Lambert-Eaton syndrome)
* A history of an anaphylactic response to Botulinum toxin type A and other involved ingredients of Investigational product
* Subjects of reproductive age who do not agree to use suitable contraceptive methods for the duration of the study

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2017-07-06 (Actual); Primary Completion 2018-10-31 (Actual); Study Completion 2018-11-05 (Actual)

PRIMARY OUTCOMES:
Change in Toronto Western Spasmodic Torticollis Rating Scale Total Score From Baseline | week 4 follow-up visit

SECONDARY OUTCOMES:
Toronto Western Spasmodic Torticollis Rating Scale Severity Subscale as a change From Baseline | week 4 follow-up visit
Toronto Western Spasmodic Torticollis Rating Scale Disability Subscale as a change From Baseline | week 4 follow-up visit
Toronto Western Spasmodic Torticollis Rating Scale Pain Subscale as a change From Baseline | week 4 follow-up visit

CONTACTS AND LOCATIONS:
Locations (1):
- Asan Medical Center, Seoul, South Korea